CLINICAL TRIAL: NCT00634803
Title: Clinical Trial of Integrated Treatment for Pain and Opioid Dependence
Acronym: POD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0608001776; 1R01DA024695-01A2 (NIH)
Record Dates: First submitted 2008-01-02; First posted 2008-03-13 (Estimated); Results first posted 2020-09-01 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Opiate Dependence; Chronic Pain
MeSH Terms: conditions — Opioid-Related Disorders; Chronic Pain | interventions — Buprenorphine; Practice Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CBT for POD (Experimental): Integrated cognitive behavioral therapy for chronic pain and opioid dependence
  Interventions: Behavioral: CBT; Drug: Buprenorphine
- Educational Counseling for POD (Active Comparator): Educational Counseling is a didactic, lecture-discussion format to supplement the information and advice provided by physicians in physician management (PM)
  Interventions: Drug: Buprenorphine; Other: Educational Counseling
- Physician Management (Active Comparator): PM is a relatively brief intervention that approximates the medically focused advice and brief counseling about medical issues that is typically provided by physicians to patients with chronic pain or other chronic medical conditions, such as diabetes or asthma.
  Interventions: Drug: Buprenorphine; Other: Physician Management

INTERVENTIONS:
Behavioral: CBT — Cognitive behavioral therapy
  Arms: CBT for POD
Drug: Buprenorphine — buprenorphine/naloxone
Other: Educational Counseling — Didactic, lecture-discussion format to supplement information and advice provided by physicians
  Arms: Educational Counseling for POD
Other: Physician Management — Brief physician counseling
  Arms: Physician Management

SUMMARY:
This study is designed to develop an effective psychotherapy for chronic pain and opioid dependence.

DETAILED DESCRIPTION:
This study aims to develop a novel manualized intervention using tailored cognitive-behavioral treatment (CBT) and buprenorphine medication to effectively treat the co-occurring disorders of non-malignant pain and opioid dependence (POD).

Specific Aims:

1. To conduct a pre-pilot phase with 16 patients with POD receiving buprenorphine maintenance treatment (BMT). In the pre-pilot phase, we will also explore the effects of different daily buprenorphine dosages on pain and opiate use.
2. To conduct a pilot randomized, clinical trial to obtain data regarding the feasibility, acceptability and efficacy (compared to Physician Management(PM) only) of manual-guided CBT or Educational Counseling (EC) for patients with POD treated with BMT (N=75).

The secondary outcomes: Development of a Treatment Manual and Development and Modification of Initial Therapy Training and Process Rating Measures were process measures and not been to be included as measures associated with RCT. These outcomes were removed when the RCT results were entered. In addition, outcomes were renamed for clarification.

At results entry, the timeframe (16 weeks) was also corrected to account for the actual timeframe used for analysis in the study. The 16-week study period listed in the protocol included a 2-week buprenorphine induction period (before randomization) and up to a 2-week post-conclusion of the clinical trial continuation on buprenorphine and referral to continuing treatment. In prior studies with buprenorphine, the study team had observed an artificially high attrition during the last 2 weeks of the planned study protocol, when participants were attempting to transition to available clinical treatments outside of the study. Consequently, as per the original study protocol for this study, the plan was to analyze intake and induction data (as baseline data) and then the data from the first 12-weeks post-randomization.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* prescription opioid addiction criteria
* moderate to severe chronic pain
* seeking or interested in buprenorphine maintenance
* understand English

Exclusion Criteria:

* methadone maintenance at a dose greater than 40 mg daily
* current suicide or homicide risk
* life-threatening or unstable medical problem
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2009-09; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Schottenfeld, MD, Principal Investigator — Yale University
Locations (1):
- Methadone Research Unit, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Barry DT, Cutter CJ, Beitel M, Kerns RD, Liong C, Schottenfeld RS. Psychiatric Disorders Among Patients Seeking Treatment for Co-Occurring Chronic Pain and Opioid Use Disorder. J Clin Psychiatry. 2016 Oct;77(10):1413-1419. doi: 10.4088/JCP.15m09963. PMID 27574837

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CBT for POD | Educational Counseling for POD | Physician Management
Started | 30 | 30 | 30
Month 1 | 29 | 29 | 29
Month 2 | 26 | 26 | 28
Month 3 | 25 | 23 | 26
Completed | 24 | 23 | 23
Not Completed | 6 | 7 | 7
Not completed — Lost to Follow-up | 6 | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CBT for POD | Educational Counseling for POD | Physician Management | Total
Number analyzed (Participants) | 30 | 30 | 30 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 30 | 90
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.3 (9.4) | 37.0 (9.9) | 35.3 (10.00) | 35.8 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 10 | 10 | 39
  Male | 11 | 20 | 20 | 51
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 30 | 90

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity
Description: Pain intensity comprises the average of 4 items related to current pain and past-week average pain, pain at its worst, and pain at its least. Pain intensity is scored on 0-10 scale (average score ranges from 0-10), where higher scores indicate higher pain intensity.Originally labeled as Pain Reduction at 16 weeks- 3 months was the correct timeframe.
Time Frame: 3 months
Population: The analysis population is the intention to treat population and all observations across time periods were used in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBT for POD | Educational Counseling for POD | Physician Management
Number analyzed (Participants) | 30 | 30 | 30
units on a scale
  Intake/Induction | 5.43 (1.34) | 5.92 (1.57) | 5.28 (1.34)
  Month 1: number analyzed (Participants) | 29 | 29 | 29
  Month 1 | 4.75 (1.62) | 5.02 (1.45) | 4.53 (1.46)
  Month 2: number analyzed (Participants) | 26 | 26 | 28
  Month 2 | 4.79 (1.50) | 4.98 (1.76) | 4.72 (1.81)
  Month 3: number analyzed (Participants) | 25 | 23 | 26
  Month 3 | 4.41 (1.67) | 4.62 (1.91) | 4.84 (1.91)

2. Primary Outcome: Number of Opioid-negative Urine Toxicology Tests
Description: Reduced illicit opioid use is defined as the number of documented opioid negative urine tests in each of the time periods.This measures the reduction in illicit opioid use - more opioid-negative tests means greater reductions in illicit opioid use. The highest possible score is 4- which would indicate 4 negative urine tests during the assessment period. Originally titled "Reduced illicit opioid use" and the timeframe was listed as 16 weeks.
Time Frame: 3 Months
Population: The analysis population is the intention to treat population and all observations across time periods were used in the analysis. Participants may have contributed to this outcome but were lost to follow up during the time period and were not measured on pain related outcomes.
Measure: Mean (Standard Deviation); unit: opioid negative urine tests
Arm/Group | CBT for POD | Educational Counseling for POD | Physician Management
Number analyzed (Participants) | 30 | 30 | 30
opioid negative urine tests
  Intake/Induction | 0.67 (0.55) | 0.67 (0.48) | 0.55 (0.69)
  Month 1: number analyzed (Participants) | 29 | 29 | 29
  Month 1 | 2.67 (1.42) | 2.80 (1.27) | 2.48 (1.70)
  Month 2: number analyzed (Participants) | 26 | 26 | 28
  Month 2 | 2.96 (1.48) | 3.30 (1.14) | 2.56 (1.72)
  Month 3: number analyzed (Participants) | 25 | 23 | 26
  Month 3 | 2.80 (1.38) | 3.25 (1.22) | 2.04 (1.71)

3. Primary Outcome: Pain Interference
Description: Pain interference comprises the average of 7 items related to past-week pain-related interference in general activity, walking, work, mood, enjoyment of life, relations with others, and sleep. Each item is scored on a 0-10 scale (averaged 0-10), where higher scores indicate higher pain interference.
Time Frame: 3 Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBT for POD | Educational Counseling for POD | Physician Management
Number analyzed (Participants) | 30 | 30 | 30
units on a scale
  Intake/Induction | 5.75 (2.12) | 5.48 (2.23) | 5.01 (2.19)
  Month 1: number analyzed (Participants) | 29 | 29 | 29
  Month 1 | 4.15 (2.09) | 3.74 (1.82) | 3.32 (2.12)
  Month 2: number analyzed (Participants) | 26 | 26 | 28
  Month 2 | 4.08 (2.06) | 3.61 (1.97) | 3.45 (2.45)
  Month 3: number analyzed (Participants) | 25 | 23 | 26
  Month 3 | 3.22 (1.94) | 3.23 (2.27) | 3.87 (2.56)

ADVERSE EVENTS:
Time Frame: Up to the end of study (month 3)
Arm/Group | CBT for POD | Educational Counseling for POD | Physician Management
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No